CLINICAL TRIAL: NCT06007092
Title: Multicentric Randomized Phase I/IIa Trial of the Safety and Immunogenicity of a Therapeutic Anti-HPV DC Targeting Vaccine in Patients With Human Papillomavirus (HPV)-Positive Oropharyngeal Cancer
Brief Title: Therapeutic Vaccine in Patients With Human Papillomavirus HPV-positive Oropharyngeal Cancer
Acronym: HPVDCVax
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Collaborators: LinKinVax (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 2022-502930-25-00; 2022/3459 (Other: CSET number)
Record Dates: First submitted 2023-08-02; First posted 2023-08-23 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Head and Neck Carcinoma; Adult Disease
MeSH Terms: conditions — Disease

STUDY DESIGN:
Intervention Model Description: Within each group, patients will be randomized between poly-ICLC- adjuvanted CD40HVac or placebo in a 5:1 ratio.
  12 patients will be treated at each dose level (10 with vaccine and 2 with placebo).
  The patients will receive three subcutaneous injections of a poly-ICLC- adjuvanted CD40HVac or placebo:
  * The first injection will occur at week 0
  * The second injection will occur at week 4 (±7 days)
  * The third injection will occur at week 24 (±7 days)
Who Masked: Participant, Investigator
Masking Description: double blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- level dose 1 HPVDC injection (Experimental): 10 patients with experimental injection at 1.0 mg
  Interventions: Biological: HPVDC injection level dose 1
- level dose 1 placebo injection (Placebo Comparator): 2 patients with experimental injection at 1.0 mg
  Interventions: Biological: placebo injection level dose 1
- level dose 2 HPVDC injection (Experimental): 10 patients with experimental injection at 3.0 mg
  Interventions: Biological: HPVDC injection level dose 2
- level dose 2 placebo injection (Placebo Comparator): 2 patients with experimental injection at 3.0 mg
  Interventions: Biological: placebo injection level dose 2

INTERVENTIONS:
Biological: HPVDC injection level dose 1 — patient receive 3 injections of vaccine at the same level dose
  Arms: level dose 1 HPVDC injection
Biological: placebo injection level dose 1 — patient receive 3 injections of vaccine at the same level dose
  Arms: level dose 1 placebo injection
Biological: HPVDC injection level dose 2 — patient receive 3 injections of vaccine at the same level dose
  Arms: level dose 2 HPVDC injection
Biological: placebo injection level dose 2 — patient receive 3 injections of vaccine at the same level dose
  Arms: level dose 2 placebo injection

SUMMARY:
This study is a multicentric double-blind placebo-controlled dose escalation trial of a CD40HVac vaccine (humanized anti-CD40 mAb fused to HPV16 E6/E7 oncoproteins) adjuvanted with poly-ICLC (Hiltonol) in patients with HPV16 oropharyngeal carcinoma with no evidence of residual or recurrent disease after surgery and/or radiochemotherapy.

The primary objective is to determine the recommended phase 2 dose (RP2D) of a poly-ICLC(Hiltonol)-adjuvanted CD40HVac vaccine according to the safety and the capacity to elicit immune responses of different doses Two dose levels of poly-ICLC-adjuvanted CD40.HVac will be explored

* 1st dose level: CD40.HVac 1.0 mg, with 1.0 mg poly-ICLC
* 2nd dose level: CD40.HVac 3.0 mg, with 1.0 mg poly-ICLC The safety data will be reviewed by an IDSMB that will give recommendations.

DETAILED DESCRIPTION:
This study is a multicentric double-blind placebo-controlled dose escalation trial of a CD40HVac vaccine (humanized anti-CD40 mAb fused to HPV16 E6/E7 oncoproteins) adjuvanted with poly-ICLC (Hiltonol) in patients with HPV16 oropharyngeal carcinoma with no evidence of residual or recurrent disease after surgery and/or radiochemotherapy.

The primary objective is to determine the recommended phase 2 dose (RP2D) of a poly-ICLC(Hiltonol)-adjuvanted CD40HVac vaccine according to the safety and the capacity to elicit immune responses of different doses Two dose levels of poly-ICLC-adjuvanted CD40.HVac will be explored

* 1st dose level: CD40.HVac 1.0 mg, with 1.0 mg poly-ICLC
* 2nd dose level: CD40.HVac 3.0 mg, with 1.0 mg poly-ICLC The safety data will be reviewed by an IDSMB that will give recommendations. Within each group, patients will be randomized between poly-ICLC- adjuvanted CD40HVac or placebo in a 5:1 ratio.

  12 patients will be treated at each dose level (10 with vaccine and 2 with placebo).

The patients will receive three subcutaneous injections of a poly-ICLC- adjuvanted CD40HVac or placebo:

* The first injection will occur at week 0
* The second injection will occur at week 4 (±7 days)
* The third injection will occur at week 24 (±7 days) Within each dose group, a period of 7 days must be observed between the first administration of vaccine of the first patient of the group and the first administration of vaccine/placebo of the second patient of the group.

A safety monitoring is planned in each dose level group:

* If a grade 5 AE occurs (except if related to cancer) at any time, all vaccinations will be halted, inclusions in the trial will be suspended and an IDSMB meeting convened for evaluation
* If a grade 4 AE related to vaccine occurs at any time, inclusions in the trial will be suspended and an IDSMB meeting convened for evaluation
* If a grade 3 AE related to vaccine occurs at any time and does not resolve or decrease to grade 1 or baseline after 7 days, inclusions in the trial will be suspended and an IDSMB meeting convened for evaluation The IDSMB recommendations as to whether or not to continue the trial after its assessment of the AE will be transmitted to the Steering Committee and to the sponsor.

Enrolment into the second dose group will open depending on the safety data of the first dose group during the safety observation period and after IDSMB and Steering Committee validation. For each patient, this safety observation period begins from the first administration and stops 2 weeks after the second injection, i.e. at Week 6.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ≥ 18 years of age.
2. Willing and able to comply with scheduled visits, treatment schedule, laboratory testing, and other requirements of the study.
3. Subjects with histologically confirmed oropharyngeal squamous cell carcinoma.
4. HPV16 genotyping determined by a specified central reference laboratory with an established polymerase chain reaction (PCR)- based assay on FFPE archived tumor biopsies (or 10 slices of 5µm).If local HPV16 genotype assessment has been performed, the subject can be enrolled if the result shows HPV16 positivity. Confirmation of HPV16 positive status will be performed retrospectively by the central laboratory on archived tissue. Formalin- fixed tumour biopsies or surgical piece before local radical treatment can be optionally available for translational research.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
6. Comprehensive curative treatment according to the disease stage and national guidelines, completed at least 16 weeks prior to study drug administration. The recommended duration between end of curative treatment and study drug administration is 18 to 20 weeks.
7. No evidence of residual or recurrent disease on the last assessment, comprising a physical examination, a head and neck CT-scan or a head and neck MRI, and a thoracic CT Scan (and TEP-scan only for patients traited by radiotherapy or radiochemotherapy without surgery).
8. Vaccination for Covid and Flu vaccines are authorised 4 weeks before or after the administration of poly-ICLC-adjuvanted CD40HVac (2 weeks during flu period for the Flu vaccine)
9. Screening laboratory values must meet the following criteria and should be obtained within 14 days prior to randomization:

   i) White blood cell count (WBC) ≥ 2 x 109/L ii) Absolute neutrophil count (ANC) ≥ 1.5 x 109/L iii) Platelets ≥ 100 x 109/L iv) Hemoglobin ≥ 9.0 g/dL v) Serum creatinine ≤ 1.5 x upper limit of normal (ULN) or creatinine clearance (CrCl) > 40 mL/min (using the Cockcroft-Gault formula): Female CrCl = (140 - age in years) x weight in kg x 0.85/ 72 x serum creatinine in mg/dL Male CrCl = (140 - age in years) x weight in kg x 1.00 / 72 x serum creatinine in mg/dL vi) Hepatic function: Total bilirubin ≤ 1.5 x ULN. Subjects with Gilbert's Disease and total bilirubin up to 3 x ULN may be eligible if total bilirubin< 3.0 mg/dL.Transaminases (ALT and AST) ≤ 3 x ULN, Alkaline phosphatase ≤ 2.5 x ULN
10. Participants who were born female: negative serum or urine beta human chorionic gonadotropin (β-HCG) pregnancy test performed before randomisation and on the day of initial IMP administration (W0)

    • Reproductive status: if heterosexually active female, consistently using an effective method of contraception with partner for sexual activity that could lead to pregnancy from at least 21 days prior to enrolment through 4 months after the last administration.

    Effective contraception is defined as using any of the following methods:
    * Condoms (male or female) with or without a spermicide;
    * Intrauterine device (IUD);
    * Intrauterine hormone releasing system (IUS);
    * Hormonal contraception (progesterone only);
    * Successful vasectomy in the male partner (considered successful if a participant reports that a male partner has (i) documentation of azoospermia by microscopy, or (ii) a vasectomy more than 2 years ago with no resultant pregnancy despite unprotected sexual activity postvasectomy);
    * Or not be of reproductive potential, such as having reached menopause (no menses for 1 year without an alternative medical cause) or having undergone hysterectomy, bilateral oophorectomy, or tubal ligation.
    * Agree not to seek pregnancy including through alternative methods, such as artificial insemination or in vitro fertilization until 4 months after the last administration.

    Participants who were born male, if heterosexually active male, using an effective method of contraception with their partner from the first day of IMP administration until 4 months after the last administration. This also applies to sperm donation.
11. Patient should understand, sign, and date the written informed consent form prior to any protocol-specific procedures performed.
12. Patients must be affiliated to a social security system or beneficiary of the same

Exclusion Criteria:

1. Clinical evidence on physical or radiological examination of residual or recurrent HPV-driven carcinoma on the primary site, in neck lymph nodes, or in any distant site metastasis.
2. Any serious or uncontrolled medical disorder that, in the opinion of the investigator, may increase the risk associated with study participation or study drug administration, impair the ability of the subject to receive protocol therapy, or interfere with the interpretation of study results.
3. Subjects with active, known, diagnosed or suspected auto-immune disease. Subjects suffering from vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune thyroiditis only requiring thyroid hormone replacement therapy, or psoriasis not requiring systemic treatment can be enrolled.
4. Patients diagnosed with active interstitial lung disease (ILD)/pneumonitis or a history of ILD/pneumonitis within the last 5 years, or another condition requiring immunosuppressive doses of medication such as systemic corticosteroids or absorbed topical corticosteroids (doses ≥ 10 mg/day prednisone or equivalent) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical corticosteroids and adrenal replacement doses < 10 mg daily prednisone or equivalent are permitted.
5. Subjects requiring maintenance treatment with immunosuppressive doses of systemic corticosteroids. Subjects being treated with a short course of corticosteroids (> 10 mg/day prednisone equivalents) should discontinue this therapy at least 2 weeks prior to start of study treatment.
6. Prior treatment with therapeutic anti-HPV vaccines.
7. Invasive surgery (defined as surgical intervention requiring general or spinal anesthesia, and hospital admission) within 28 days prior to start of study treatment.
8. Uncontrolled infection with human immunodeficiency virus (HIV), hepatitis B virus or hepatitis C virus.
9. Patient with active infection must be postponed until infection resolution
10. Subjects with an uncontrolled or significant heart disease such as long QT syndrome with QTcF > 480 ms on baseline ECG, NYHA III/IV or uncontrolled arrhythmia.
11. History of organ transplantation, including allogenic peripheral stem cell or bone marrow transplantation.
12. Participation in another clinical study with an investigational product during the last 6 months and while on study treatment
13. Vaccination for Covid and Flu vaccines is not permitted within 4 weeks prior the first vaccination with polyICLC adjuvanted CD40HPVac (2 weeks during flu period for the Flu vaccine.
14. Treatment is not permitted within 4 weeks prior the first vaccination and 4 months after the last injection. Furthermore, the use of this medication will be considered as a deviation to the protocol.

    * curative treatment within 12 weeks before the first injection,
    * Corticosteroids,
    * Live attenuated vaccines (such as measles, mumps, and rubella [MMR]; oral polio vaccine [OPV]; varicella; yellow fever) or any vaccines that are not live attenuated (eg, tetanus, pneumococcal, Hepatitis A or B) except IMP vaccine.
    * Immunosuppressive medications (Not excluded: [1] corticosteroid nasal spray; [2] inhaled corticosteroids; [3] topical corticosteroids for mild, uncomplicated dermatitis; or [4] a single course of oral/parenteral corticosteroids at doses < 2 mg/kg/day and length of therapy < 11 days with completion at least 30 days prior to enrollment)
    * Blood products
    * Immunoglobin
    * Anti-tuberculosis drugs
    * Immunomodulators (such as cytokines or interferons) or immunosuppressive drugs during 8 weeks preceding the screening visit and as of 4 months after the last injection will not be allowed. If any patient needs chronic use of one of these medicine during this period, the subject will be withdrawn from the investigational product but should be followed at all visits as planned by the protocol
    * Antipyretic will not be allowed twelve (12) hours before immunization as preventive treatment of pain or fever.
15. Pregnant or breastfeeding women or intending to become pregnant during study
16. Patient under guardianship or deprived of his liberty by a judicial or administrative decision or incapable of giving its consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-07-31 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
immunological outcomes: The frequency (%) of HPV16-specific T cells | at the end of the study, 24 months after the first inclusion
  The primary immunological outcomes is: The frequency (%) of HPV16-specific T cells will be evaluated using Activation Induced Marker (AIM) assay using CD69 and CD137 (4-1BB) activation markers after a 24 hours stimulation using two validated tests routinely used in vaccine studies including ICS and AIM assays. These tests will be performed in all collected samples at W0, W2, W6, W26 and W48 for the durability of the responses.
recommended phase 2 dose (mg) (RP2D) of poly-ICLC-adjuvanted CD40HVac | 1year after the last visit of last patient
  The recommended phase 2 dose (RP2D) of poly-ICLC-adjuvanted CD40HVac will be determined by the Extensive Steering Committee according to the safety analysis and to the capacity of the vaccine to elicit immune responses. The capacity to elicit immune response will be used to choose the RP2D in the event that several doses of vaccine are acceptable in terms of safety (i.e. that meet of the "go-criterion").

CONTACTS AND LOCATIONS:
Overall Officials: Caroline EVEN, Dr, Study Chair — Gustave Roussy, Cancer Campus, Grand Paris
Locations (1):
- Gustave Roussy, Villejuif, France

IPD SHARING:
Plan to Share IPD: No